CLINICAL TRIAL: NCT00967811
Title: An Open-Label, Phase 2 Study of Different Formulations (E1 and E2) of the Latanoprost Punctal Plug Delivery System (L-PPDS) in Subjects With Ocular Hypertension (OH) or Open-Angle Glaucoma (OAG)
Brief Title: A Study of Different Formulations of the L-PPDS in Subjects With OH or OAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPL GLAU 07
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Formulation E1 (Experimental): Formulation E1 of Latanoprost-PPDS
  Interventions: Drug: Formulation E1 of L-PPDS
- 2. Formulation E2 (Experimental): Formulation E2 of Latanoprost-PPDS
  Interventions: Drug: Formulation E2 of L-PPDS

INTERVENTIONS:
Drug: Formulation E1 of L-PPDS — Control of IOP compared to baseline for Formulation E1 of the experimental dose of Latanoprost-PPDS for 6 weeks or until loss of efficacy.
  Arms: 1. Formulation E1
Drug: Formulation E2 of L-PPDS — Control of IOP compared to baseline for Formulation E2 of experimental dose of Latanoprost-PPDS for 6 weeks or until loss of efficacy.
  Arms: 2. Formulation E2

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of two formulations of the Latanoprost-PPDS in subjects with ocular hypertension or open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age diagnosed with ocular hypertension or open-angle glaucoma
* Subjects who have a best corrected visual acuity of 20/100 or better

Exclusion Criteria:

* Subjects who wear contact lenses
* Subjects who have uncontrolled medical conditions
* Subjects requiring chronic topical artificial tears, lubricants, and/or requiring any other chronic ocular topical medications
* Subjects who have a history of chronic or recurrent inflammatory eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
IOP change from baseline | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Cuzzani, MD, Study Director — QLT Inc.
Locations (1):
- Menlo Park, California, United States